CLINICAL TRIAL: NCT04796727
Title: ONe Year Follow-up in Patients Admitted for Emergency Coronary Angiography After Rescuscited Cardiac Arrest
Brief Title: One Year Follow-up After Rescuscited Cardiac Arrest
Acronym: ONYRCA
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0285
Record Dates: First submitted 2021-02-25; First posted 2021-03-15 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Cardiac Arrest
Keywords: neurological state; Cardiological state; Quality of life; Coronary angiography; One year mortality; Cardiac vents; One year quality of life; Neurological events
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OHCA: 300 OHCA admitted directly to the cathlab and alive at discharge during a 2 years period of enrolement.

SUMMARY:
While 80 % of all sudden cardiac death (SCD) result from coronary artery disease (CHD) approximatively 2/3 of SCD occur as a first manifestation of the CHD. VF (ventricular fibrillation) is the main cause of SCD in acute coronary syndrome (ACS), and the 2017 ESC Guidelines for the management of acute myocardial infarction, recommended direct admission to the catheterization laboratory in survivors of out of hospital cardiac arrest (OHCA) with criteria for STEMI on the post-resuscitation electrocardiogram (ECG) (Class I, grade B). However, During the past few years, the number of immediate coronary angiography (CA) for suspected ACS in patients presenting an OHCA increased, with a survival rate at discharge in this subgroup of patients better, about 60 to 80% (1). However, the survival rate remains poor in the global population of OHCA and some survivors patients may have neurological sequelles, related to global anoxia consequences or altered quality of life related to cardiac function impairement .

While the survival rate at hospital discharge is well known, the investigators have few data on long term outcomes , particularly regarding cardiac and neurological states.

Therefore the main objective of this study is to evaluate prospectively, in an observational study, the one-year prognosis of patients with rescuscited OHCA in whom a CA for suspected ACS was performed in the university hospital of Montpellier. Only patients alive at discharged are considered for the follow-up to eliminate the in-hospital mortality .

The investigators aim to assess year neurological status using medical questionnaires at one year follow-up(primary end point). The investigators hypothesize that 10% of patients will discharged alive from hospital with severe neurological sequelae at 1 year.Secondary end point will evaluate cardiac status, quality of life and pronostic factors of adverse outcome.

DETAILED DESCRIPTION:
Patients older than 18 years old undergoing CA for cardiac arrest discharged alive from hospital will be included from January 1, 2018 to May 31, 2020.

The investigators exclude all the patients who died during the in-hospital stay and patients who had VF immediately rescucitated by electric cardioversion including only unconscious patients at admission in the cath lab. Patients were also excluded if they did not receive active in-hospital treatment after cardiac arrest based on either a do-not-attempt-resuscitation order, end-stage malignancy preceding the arrest, or had minimal chances of meaningful survival (defined as not witnessed cardiac arrest with asystole, lengthy resuscitation, or advanced age).

Patient characteristics, modalities of cardiac arrest and intra-hospital progress were collected using DxCare software.

Cardiac and neurological status will be collected at 1 year follow-up either by using consultation report or by a phone call If available, an initial evaluation is done at 3 months.

Cerebral Performance Category (CPC) will be used to assess the neurological functional status Primary end point is the rate of patients with severe neurological sequelae at one year follow-up defined as CPC category ≥ 3.

Secondary ends points will evaluate the survival rate, NYHA functional class, rehospitalization and quality of life at 1 year.

Quality of life at one year is recorded using the QOLIBRI (Quality of Life after Brain Injury) which is a novel health-related quality-of-life (HRQoL) instrument specifically developed for traumatic brain injury (TBI) (2). It provides a profile of HRQoL in six domains together with an overall score. The questionnaire is completed by asking questions by phone to patients available at 1 year follow-up.

The inclusion of 96 patients will make possible to highlight a frequency of severe neurological sequelae of 10 percent with a precision of 5 percent (width of the confidence interval) and considering an alpha risk of 5 percent.

Considering that our active patient file include 150 cardiac arrests per year, of which 50 are discharged alive per year, the inclusion of 96 patients discharged alive from hospital over a 2-year period seems to be realistic.

ELIGIBILITY:
Inclusion criteria:

* Older than 18 years old.
* Out of Hospital Cardiac arrest
* Coronary angiography in emergency
* Alive at discharge.

Exclusion criteria:

* Absence of return of spontaneous circulation after reanimation.
* Admission in a resuscitation unit before the coronary angiography.
* In-hospital death.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 who are admitted directly to our cath lab for a cardiopulmonary arrest and alive at discharge.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Incidence of patients alive without neurological sequelae | 1 year
  Incidence of patients alive without neurological sequelae at one year follow up after out of hospital cardiac arrest. Neurological status will be evaluated with the Cerebral Performance Category score. Patients with a score of 1 or 2 will be considered without neurological sequelae. Grade 1 correspond to patients with normal cerebral performance and grade 2 to patients with moderate cerebral disability but don't need any support for daily activities. Grade 3 is for patients with severe disability leading to daily support. Grade 4 is for coma or vegetative state and Grade 5 for brain death.
Incidence of patients alive | 3 months
  Incidence of patients alive Incidence of patients alive without neurological sequelae (CPC 1 or 2)
Incidence of patients alive | 1 year
  Incidence of patients alive Incidence of patients alive without neurological sequelae (CPC 1 or 2)
Rate of hospitalizations | 1 year
  Rate of hospitalizations (from cardiovascular cause)
Rate of hospitalizations | 3 months
  Rate of hospitalizations (from cardiovascular cause)

SECONDARY OUTCOMES:
Cardiac functional status | 1 year
  Cardiac functional status using the NYHA scale (1 or 2 for good functional status)
Cardiac functional status | 3 months
  Cardiac functional status using the NYHA scale (1 or 2 for good functional status)

CONTACTS AND LOCATIONS:
Overall Officials: Florence Leclercq, PU PH, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Result] Patel N, Patel NJ, Macon CJ, Thakkar B, Desai M, Rengifo-Moreno P, Alfonso CE, Myerburg RJ, Bhatt DL, Cohen MG. Trends and Outcomes of Coronary Angiography and Percutaneous Coronary Intervention After Out-of-Hospital Cardiac Arrest Associated With Ventricular Fibrillation or Pulseless Ventricular Tachycardia. JAMA Cardiol. 2016 Nov 1;1(8):890-899. doi: 10.1001/jamacardio.2016.2860. PMID 27627616
- [Result] von Steinbuchel N, Wilson L, Gibbons H, Hawthorne G, Hofer S, Schmidt S, Bullinger M, Maas A, Neugebauer E, Powell J, von Wild K, Zitnay G, Bakx W, Christensen AL, Koskinen S, Formisano R, Saarajuri J, Sasse N, Truelle JL; QOLIBRI Task Force. Quality of Life after Brain Injury (QOLIBRI): scale validity and correlates of quality of life. J Neurotrauma. 2010 Jul;27(7):1157-65. doi: 10.1089/neu.2009.1077. PMID 20210602